CLINICAL TRIAL: NCT02361619
Title: An Open-label Crossover Trial Assessing the Value of Dabigatran in a Drug Interaction Cocktail in Healthy Young Volunteers
Brief Title: Dabigatran in an Interaction Probe Drug Cocktail
Acronym: D-cocktail
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: T162/2014; 2014-003628-38 (EudraCT Number)
Record Dates: First submitted 2015-01-30; First posted 2015-02-12 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Caffeine; Diclofenac; Esomeprazole; Metoprolol; Midazolam; Dabigatran; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Caffeine; Drug: Diclofenac; Drug: Esomeprazole; Drug: Metoprolol; Drug: Midazolam; Drug: Dabigatran; Drug: Clarithromycin

INTERVENTIONS:
Drug: Caffeine — probe
Drug: Diclofenac — probe
Drug: Esomeprazole — probe
Drug: Metoprolol — probe
Drug: Midazolam — probe
Drug: Dabigatran — probe
Drug: Clarithromycin — perpetrator

SUMMARY:
Four periods of oral dosing following overnight fasting (1. known metabolic probe drug cocktail consisting of caffeine, diclofenac, esomeprazole, metoprolol, midazolam; 2. dabigatran + cocktail; 3. dabigatran alone; 4. clarithromycin 3 days + cocktail + dabigatran). Blood samples collected for pharmacokinetics over 24 h. Washout between periods. Adverse events, haematology and clinical chemistry recorded.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Weight at least 50 kg and body mass index 19 - 30 kg m-2
* Normal clinical laboratory profiles
* No childbearing potential or use of adequate contraceptive measures

Exclusion Criteria:

* Blood loss >300 ml within 2 months prior to the first dosing day
* Pregnancy, breastfeeding
* Allergy or hypersensitivity to caffeine, diclofenac, esomeprazole, metoprolol, midazolam, dabigatran or clarithromycin or to excipients in the pharmaceutical products
* Infection with HIV, HBV or HCV
* Participation in the preceding 3 months or concomitantly in any clinical drug study
* Suspected current drug or alcohol abuse
* History of drug or alcohol abuse.
* Concomitant medication with the exception of hormonal contraception.
* Positive result in urine test for drug abuse.
* Nicotine consumption equivalent to >5 cigarettes per day

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-02; Primary Completion 2016-09 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
AUC of dabigatran in plasma | 24 h
  Exposure ratio for dabigatran in combination and dabigatran alone

SECONDARY OUTCOMES:
Number of subjects with adverse events | 23 days

CONTACTS AND LOCATIONS:
Overall Officials: Petri Vainio, MD PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Teutori CPRU, Turku, Finland